CLINICAL TRIAL: NCT00391287
Title: A Prospective, Immunogenicity Surveillance Registry (PRIMS) to Estimate the Incidence of Erythropoietin Antibody-Mediated Pure Red Cell Aplasia Among Subjects With Chronic Renal Failure and Subcutaneous Exposure to Recombinant Erythropoietin Products
Brief Title: Surveillance Study to Estimate the Incidence of Pure Red Blood Cell Aplasia Among Patients With Chronic Kidney Failure
Acronym: PRIMS
Status: Completed | Type: Observational
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Collaborators: Janssen-Cilag International NV (Industry)
Responsible Party: Sponsor
Other Study IDs: CR011587; EPOANE4014 (Other: Janssen-Cilag International NV); 001992-001 (Other: Legacy System ID)
Record Dates: First submitted 2006-10-20; First posted 2006-10-23 (Estimated); Last update posted 2014-10-03 (Estimated); Status verified 2014-10

CONDITIONS: Pure Red-Cell Aplasia; Chronic Kidney Failure
Keywords: Red-Cell Aplasia due to Chronic Kidney Failure; Aplastic Anemia; Recombinant Erythropoietin; Surveillance Registry; Registries
MeSH Terms: conditions — Red-Cell Aplasia, Pure; Kidney Failure, Chronic; Anemia, Aplastic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- erythropoietin treatment in CRF: Patients exposed to EPREX or other marketed erythropoietin products administered by the subcutaneous route of administration for the treatment of anemia of Chronic Renal Failure

SUMMARY:
The purpose of this study is to estimate the incidence rate of pure red cell aplasia (PRCA; aplastic anemia) mediated by erythropoietin (EPO) antibodies in patients who are receiving subcutaneous (s.c.) epoetin alfa (polysorbate 80 formulation) for the treatment of anemia associated with chronic renal failure (CRF), and to compare this incidence rate to the incidence rate with s.c. exposure to other currently marketed recombinant erythropoietin products (epoetin alfa, epoetin beta, darbepoetin alfa), with adjustment of duration for which the drug is given to the patient. The study will also examine the impact of the pattern of using mixed s.c. exposure to multiple erythropoietin products occurring in this patients, and the impact of the time from which the treatment is started to the onset of PRCA.

DETAILED DESCRIPTION:
In 1998, prompted by concern that human serum albumin (HAS- the stabilizer in the epoetin alfa formulation) could theoretically transmit Creutzfeldt-Jakob disease and bovine spongiform encephalopathy, an alternative epoetin alfa formulation using polysorbate 80 as a stabilizer was introduced. The polysorbate 80 epoetin alfa formulation became available in a variety of product presentations (i.e., single-use vials and prefilled syringes with both coated and uncoated stoppers) to provide for prescribing flexibility, patient convenience, and choice of route of administration. Soon after the introduction of the polysorbate 80 epoetin alfa formulation in prefilled syringes, an increasing number of cases of EPO antibody-mediated pure red cell aplasia (PRCA) were reported in patients with chronic renal failure (CRF) exposed to epoetin alfa by the s.c. route. This led to contraindication of the s.c. route for epoetin alfa in the European Union (E.U.) and Switzerland in December 2002. It was subsequently shown that the increased risk for PRCA was associated with one specific polysorbate 80 epoetin alfa presentation - prefilled syringes with uncoated rubber stoppers. It appeared that uncoated rubber stoppers, when exposed to polysorbate 80, released organic compounds (leachates) into the epoetin alfa formulation, and that these leachates were the most probable product-specific cause for the increase in EPO antibody-mediated PRCA. A worldwide recall of the polysorbate 80 epoetin formulation in prefilled syringes with uncoated stoppers was completed in March 2004. FluroTec-coated stoppers are now used in all prefilled syringes containing the polysorbate 80 epoetin alfa formulation, to prevent leachates from entering the formulation. Following these actions, the incidence rate of EPO antibody-mediated PRCA in CRF patients receiving s.c. epoetin alfa fell to a level similar to that for the HSA-containing epoetin formulation, which has a long-standing and well-characterized safety profile. As of 30 November 2005, s.c. exposure in CRF patients to the polysorbate 80 epoetin alfa formulation in prefilled syringes with coated stoppers was 71,880 patient-years, with 4 cases of EPO antibody-mediated PRCA reported. In 2006, E.U. Health Authorities reauthorized s.c. epoetin alfa use in CRF patients for whom intravenous access is not readily available. As part of the reauthorization, the sponsor agreed to conduct this registry in order to demonstrate that the polysorbate 80 epoetin alfa formulation using a coated stopper has an acceptable immunogenic safety profile and to define the incidence of EPO antibody-mediated PRCA associated with recombinant erythropoietin use among patients with anemia associated with CRF. This is a multicenter, multinational, immunogenicity surveillance registry using a prospective cohort design (patients identified by a common characteristic), with enrollment of parallel groups that are exposed to the polysorbate 80 formulation of epeotin alfa or other marketed erythropoietin products administered by the s.c. route of administration for the treatment of anemia associated with CRF. The registry is designed to address the following question: Is the current rate of PRCA with the s.c. polysorbate 80 epoetin alfa formulation using coated stoppers similar to the current rate with other marketed erythropoietin products administered by the s.c. route, adjusted for duration of exposure? Each patient will be observed for development of PRCA for up to 3 years. Information on exposure to erythropoietin products, stage of CRF, treatment modality for CRF, erythropoietin handling and storage information, and most recent hemoglobin level will be collected quarterly. Cases of unexplained loss or lack of effect (LOE) with an administered erythropoietin product, including cases of suspected PRCA, will be reported to the sponsor as serious adverse events. Cases of EPO antibody-mediated PRCA will be determined by the clinical presence of suspected PRCA, an unexplained LOE with administered erythropoietin product, and the presence of EPO antibody. An Independent Case Adjudication Committee will review blinded case data for patients with unexplained LOE and identify cases of EPO antibody-mediated PRCA. A separate Independent Safety Advisory Committee will be responsible for periodically reviewing unblinded patient data and summary data and will make recommendations related to the incidence rate of PRCA associated with s.c. epoetin alfa use. The sponsor will actively monitor registry enrollment and erythropoietin brand usage to ensure that the registry accrues 20,000 person-years of s.c. exposure to epoetin alfa and 20,000 person-years of s.c. exposure to all other erythropoietin products combined. If it appears that one registry arm will meet this accrual goal before the other, the sponsor may elect to selectively close those investigational sites with predominant use of the erythropoietin product(s) in the arm approaching full accrual. The registry will provide no inducement to change therapy and will be non-interventional.

ELIGIBILITY:
Inclusion Criteria:

* Patients with established CRF as an indication for the treatment of anemia
* Patients who are receiving or are about to receive (within 1 month) a marketed erythropoietin (i.e., epoetin alfa [EPREX/ERYPO/GLOBUREN], epoetin beta [NEORECORMON®], or darbepoetin alfa [ARANESP®]) by the s.c. route of administration
* Patients who are likely to continue to receive s.c. erythropoietin product(s) for at least 1 year.

Exclusion Criteria:

* Patients with a history of pure red cell aplasia or aplastic anemia
* Patients who are experiencing unexplained loss or lack of effect to a recombinant erythropoietin product ongoing at the time of enrollment
* Patients who have had prior recombinant erythropoietin treatment whose anemia had never responded (primary lack of efficacy)
* Patients with a history of EPO antibodies prior to enrollment
* Subjects who are currently receiving immunosuppressive medication (e.g., cyclosporine, tacrolimus, sirolimus, mycophenolic mofetil, azathioprine, or monoclonal antibodies) or corticosteroids at a dose corresponding to >15 mg/day prednisolone
* Subjects whose first s.c. exposure to any erythropoietin product was >1 year prior to enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients should have documented chronic renal failure (CRF) and be receiving or about to receive (within 1 month) a marketed erythropoietin product by the subcutaneous route of administration at the time of enrollment. Patients may be at any stage of CRF (Stages 1 to 5) or be receiving any treatment for CRF, including predialysis, peritoneal dialysis, or hemodialysis, but should not be receiving immunosuppressive treatment following an organ transplant.
  Patients will be enrolled at sites located in the E.U. and Australia.
Sampling Method: Probability Sample
Enrollment: 15334 (Actual)
Dates: Start 2006-06; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
estimate the incidence rate of EPO antibody-mediated Pure Red Cell Aplasia (PRCA) | Unexplained Loss of Effect (LOE) follow-up
  estimate the incidence rate of EPO antibody-mediated PRCA with s.c. exposure to the polysorbate 80 formulation of epoetin alfa and to compare this incidence rate to the incidence rate with s.c. exposure to other currently marketed recombinant erythropoietin products (epoetin alfa, epoetin beta, darbepoetin alfa) with adjustment for duration of exposure.

SECONDARY OUTCOMES:
sensitivity analyses | Unexplained Loss of Effect (LOE) follow-up
  to examine, in sensitivity analyses of the incidence rates of EPO antibody-mediated Pure Red Cell Aplasia (PRCA) and their rate ratios, the impact of the patterns of mixed s.c. exposure to multiple erythropoietin products occurring in this subject population and of varying the assumption of 1 to 12 months for latency from exposure to the onset of PRCA

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.
Locations (387):
- Australia (12):
  - Adelaide
  - Central Queensland M C
  - Fremantle
  - Hobart
  - Launceston
  - Liverpool
  - Newcastle
  - Parkville
  - Perth
  - Randwick
  - Wollongong
  - Woodville
- Belgium (31):
  - Aalst
  - Antwerp
  - Arlon
  - Assebroek
  - Ath
  - Bonheiden
  - Bruges
  - Brussels
  - Charleroi
  - Deinze
  - Edegem
  - Eeklo
  - Frameries
  - Genk
  - Ghent
  - Gilly
  - Huy
  - Ieper
  - La Louvière
  - Leuven
  - Liège
  - Mons
  - Namur
  - Roeselare
  - Sint-Gillis-Dendermonde
  - Sint-Niklaas
  - St-Truiden
  - Tournai
  - Turnhout
  - Westmalle
  - Wilrijk
- Denmark (4):
  - Århus N N/A
  - Holstebro
  - Sønderborg
  - Viborg
- Finland (3):
  - Helsinki
  - Tampere
  - Turku
- Germany (184):
  - Aachen
  - Aalen
  - Altötting
  - Alzey
  - Annaberg-Buchholz
  - Ansbach
  - Arnstadt
  - Aschersleben
  - Augsburg
  - Aurich
  - Bad Bevensen
  - Bad Ems
  - Bad Homburg
  - Bad König
  - Bad Krozingen
  - Bad Mergentheim
  - Bad Nenndorf
  - Bad Oeynhausen
  - Bad Tölz
  - Bassum
  - Bergisch Gladbach
  - Berlin
  - Bernburg
  - Betzdorf
  - Biberach
  - Bielefeld
  - Bischofswerda
  - Bonn
  - Braunschweig
  - Bremen
  - Bremerhaven
  - Coburg
  - Cochem
  - Coesfeld
  - Cologne
  - Cottbus
  - Darmstadt
  - Deggendorf
  - Dillingen
  - Dinkelsbühl
  - Dormagen
  - Düsseldorf
  - Eberswalde
  - Eisenach
  - Elmshorn
  - Elsenfeld
  - Emmering
  - Emsdetten
  - Erftstadt
  - Erfurt
  - Erkelenz
  - Essen
  - Finsterwalde
  - Flensburg
  - Frankfurt
  - Freiberg
  - Freiburg im Breisgau
  - Fürstenwalde
  - Fürstenzell
  - Fürth
  - Gera
  - Göppingen
  - Greifswald
  - Gütersloh
  - Hagenow
  - Halberstadt
  - Hamburg
  - Hamelin
  - Hanover
  - Haßfurt
  - Heidenau
  - Heilbronn
  - Helmstedt
  - Herford
  - Herzberg
  - Hilden
  - Hildesheim
  - Hoyerswerda
  - Hürth
  - Ibbenbueren
  - Immenstadt im Allgäu
  - Ingolstadt
  - Jena
  - Kaiserslautern
  - Kamen
  - Kelheim
  - Kempten
  - Kerpen
  - Kiel
  - Kleve
  - Kronach
  - Kulmbach
  - Lahr
  - Landshut
  - Landstuhl
  - Langenfeld
  - Langenhagen
  - Langenselbold
  - Lehrte
  - Leipzig
  - Leverkusen
  - Lichtenfels
  - Lindau
  - Linnich
  - Lohr
  - Lübeck
  - Lüdenscheid
  - Lüneburg
  - Magdeburg
  - Malente
  - Mannheim
  - Marburg
  - Markkleeberg
  - Marl
  - Mayen
  - Meiningen
  - Moers
  - Mönchengladbach
  - Mühlhausen
  - München
  - Münster
  - Neubrandenburg
  - Neunkirchen
  - Neuruppin
  - Nuremberg
  - Nürtingen
  - Oberschleißheim
  - Offenburg
  - Olpe
  - Passau
  - Peine
  - Pfaffenhofen
  - Pforzheim
  - Potsdam
  - Quedlinburg
  - Regensburg
  - Remagen
  - Rosenheim
  - Rostock
  - Rüsselsheim am Main
  - Saarlouis
  - Sachsen
  - Saint Martin
  - Saint Wendel
  - Salzgitter
  - Schönebeck
  - Schwabach
  - Schwedt
  - Schweinfurt
  - Schwerin
  - Seehausen
  - Seelow
  - Siegen
  - Sigmaringen
  - Sindelfingen
  - Singen
  - Sinsheim
  - Sonneberg
  - Spremberg
  - Stade
  - Straubing
  - Stuttgart
  - Suhl
  - Tangermünde
  - Traunstein
  - Uelzen
  - Viersen
  - Villingen-Schwenningen
  - Waiblingen
  - Waldshut-Tiengen
  - Weinheim
  - Weißenburg
  - Weißenfels
  - Weißwasser
  - Wesseling
  - Weyhausen
  - Wiesbaden
  - Wittenberg
  - Wolfenbüttel
  - Worms
  - Wuppertal
  - Würzburg
  - Zirndorf
  - Zwickau
- Greece (15):
  - Alexandroupoli
  - Athens
  - Chalcis
  - Didimoteicho
  - Edessa
  - Grevená
  - Heraklion
  - Ioannina
  - Larissa
  - Piraias
  - Rhodes
  - Serres
  - Thessaloniki
  - Thessalonikis
  - Véroia
- Ireland (2):
  - Cork
  - Galway
- Netherlands (4):
  - 's-Hertogenbosch
  - Apeldoorn
  - Rotterdam
  - Weert
- Norway (3):
  - Oslo
  - Trondheim
  - Tvnsberg
- Poland (20):
  - Bialystok
  - Bytom
  - Chojnice
  - Ciechanów
  - Działdowo
  - Gdansk
  - Gdansk-Zaspa
  - Koszalin
  - Lodz
  - Lublin
  - Oława
  - Poznan
  - Proszowice
  - Radomsko
  - Rybnik
  - Stalowa Wola
  - Torun
  - Warsaw
  - Wroclaw
  - Łomża
- Portugal (14):
  - Aveiro
  - Barcelos
  - Braga
  - Coimbra
  - Evora
  - Faro
  - Leiria
  - P-1100 Lisboa N/A
  - Portalegre
  - Porto
  - S. Joao Da Madeira
  - Setúbal
  - Viana do Castelo
  - Vila Nova de Gaia
- Spain (20):
  - Alcorcón
  - Barcelona
  - Burgos
  - Castellon
  - Girona
  - Leganés
  - León
  - Madrid
  - Manresa
  - Marañón
  - Mollet del Vallès
  - Oviedo
  - Palma de Mallorca
  - Sabadell
  - Santa Cruz de Tenerife
  - Santander
  - Teruel
  - Valencia
  - Valladolid
  - Zaragoza
- Sweden (33):
  - Avesta
  - Bollnäs
  - Borås
  - Eksjö
  - Eskilstuna
  - Gällivare
  - Gävle
  - Gothenburg
  - Halmstad
  - Karlshamn
  - Karlskoga
  - Karlskrona
  - Köping
  - Linköping
  - Luleå
  - Malmo
  - Norrköping
  - Nyköping
  - Örebro
  - Örnsköldsvik
  - Östersund
  - Skellefteå
  - Skene
  - Skövde
  - Stockholm
  - Sundsvall
  - Trollhättan
  - Umeå
  - Uppsala
  - Varberg
  - Värnamo
  - Västerås
  - Västervik
- Switzerland (11):
  - Aarau
  - Baden
  - Bellinzona
  - Chur
  - Lausanne
  - Nyon
  - Schwyz
  - Sierre
  - Sion
  - Wil
  - Zurich
- United Kingdom (31):
  - Antrim
  - Basildon
  - Bradford
  - Brighton
  - Cambridge
  - Cardiff
  - Carshalton
  - Derby
  - Doncaster
  - Dundee
  - Edinburgh
  - Exeter
  - Great Yarmouth
  - Inverness
  - Kilmarnock
  - Leicester
  - London
  - Londonderry
  - Manchester
  - Merseyside
  - Merthyr Tydfil
  - Norwich
  - Nottingham
  - Oxford
  - Plymouth
  - Portsmouth
  - Reading
  - Sheffield
  - Shrewsbury
  - Stevenage
  - Suffolk

REFERENCES:
- See also: Prospective, Immunogenicity Surveillance Registry (PRIMS) to Estimate the Incidence of Erythropoietin Antibody-Mediated Pure Red Cell Aplasia Among Subjects With Chronic Renal Failure and Subcutaneous Exposure to Recombinant Erythropoietin Products — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=736&filename=CR011587_CSR.pdf